CLINICAL TRIAL: NCT00608036
Title: Ecological Analysis of Activity, Eating, and Weight in Adolescents
Brief Title: Evaluating the Relationship Between Physical Activity, Diet, Weight, and the Neighborhood Environment for Adolescents
Status: Completed | Type: Observational
Sponsor: Dr. James Sallis (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Dr. James Sallis, Distinguished Professor, Department Family and Preventive Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 527; R01HL083454 (NIH)
Record Dates: First submitted 2008-01-28; First posted 2008-02-06 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Obesity
Keywords: Adolescents; Neighborhood; Walkability; Physical Activity; Quality of Life; Ecological Analysis; Dietary Patterns; Weight Status; Neighborhood Environment; Food Environment; Recreation Environment
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Many teenagers have unhealthy eating habits and do not get enough physical activity. This study will examine whether the neighborhood in which a teenager lives affects his/her quality of life, physical activity levels, and eating habits.

DETAILED DESCRIPTION:
Obesity is an increasingly important health problem in the United States, particularly among adolescents. Previous studies among adults have shown that people who live in neighborhoods with good "walkability" and recreational environments have increased physical activity levels, and some studies have suggested that there is a relationship between the neighborhood food environment and eating patterns. While these concepts have been studied in adults, more research is needed on the effect of the neighborhood environment on adolescents. In this study, adolescents who live in select neighborhoods in Seattle-King County, WA and Baltimore-Washington, DC will be enrolled. Forty-eight neighborhoods in these areas will be studied, with researchers taking into account the neighborhoods' walkability levels (e.g., combination of street connectivity, residential density, land use mix, retail floor area ratio) and median income levels. Study researchers will examine and create formulas to measure walkability, pedestrian infrastructure, public recreation space, and nutrition environment quality. Researchers will also examine crime and weather patterns; psychosocial variables; parent support; and perceived neighborhood, school, and home environments. Overall, this study will evaluate the ability of a research model to explain the variation in physical activity levels, sedentary behavior, dietary patterns, and weight among adolescents, with an emphasis on neighborhood environment.

There will be no study visits for this study: participation will take place entirely through the mail, phone, or internet. Participants will include adolescents between the ages of 12 and 16 years old and their parents, all of whom live in the identified study neighborhoods. At the time of study entry, adolescents will complete a questionnaire on neighborhood and safety issues, diet, physical activity habits and places where activity occurs, grades, school policies and parental rules that affect physical activity and eating, and the support they get from people regarding healthy eating and physical activity. One parent of each adolescent will also complete a neighborhood information questionnaire. Adolescents will measure their height, weight, and waist circumference and send the measurements to study staff along with the questionnaire. Next, a 4-week period, study staff will call adolescents on three random days and collect information on their diet in the previous 24 hours. During this period, adolescents will wear an activity meter and a GPS monitor for 7 consecutive days and will mail the devices to study staff for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Child is between 12 and 16 years old
* Child and parent live in identified block group
* Child and parent speak English
* Child attends middle school or high school

Exclusion Criteria:

* Child must not have a diagnosed thought disorder, suicidality, substance abuse disorder, or other psychological or medical condition that would prevent full participation in the study
* Child must not have a disability or illness that would prevent moderate intensity physical activity
* Child must not have an eating disturbance indicative of significant eating disorder pathology

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be selected from identified neighboorhoods in the Seattle-King County, WA and Baltimore-Washington, DC areas.
Sampling Method: Probability Sample
Enrollment: 954 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Physical Activity measured with accelerometer | Time 1
  Average minutes of moderate-to-vigorous physical activity per day, average minutes of sedentary time per day

SECONDARY OUTCOMES:
Diet measured with 24 hour dietary recall interviews | Time 1
  Measures of diet quality

CONTACTS AND LOCATIONS:
Overall Officials: James F. Sallis, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - Children's Hospital and Regional Medical Center, Seattle, Washington